CLINICAL TRIAL: NCT02017210
Title: Insulin-sensitive Obesity: Prospective and Interventional Studies
Brief Title: Insulin-sensitive Obesity: Lessons From Longitudinal Data
Acronym: ISOS
Status: Completed | Type: Observational
Sponsor: Garvan Institute of Medical Research (Other)
Collaborators: The University of Hong Kong (Other); Life for a Child Program, Diabetes Australia (Other); The University of New South Wales (Other); University of Sydney (Other); St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Dorit Samocha-Bonet, Group leader Clinical Insulin Resistance Group, Garvan Institute of Medical Research
Other Study IDs: ISOS (SVH 13/143)
Record Dates: First submitted 2013-12-09; First posted 2013-12-20 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Insulin Sensitivity/Resistance; Obesity
Keywords: Hyperinsulinaemic-euglycaemic clamp; Body fat composition; Dual-energy x-ray absorptiometry; Obesity; Insulin resistance
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma, subcutaneous abdominal fat, skeletal muscle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lean/normal weight: Individuals with body mass index (BMI)<25 kg/m^2 in the baseline study
- Overweight/Obese Insulin-Sensitive: Individuals with BMI>25kg/m^2 who were deemed insulin-sensitive by the hyperinsulinemic -euglycemic clamp (with M/I value above median for men and women separately)
- Overweight/Obese Insulin-Resistant: Individuals with BMI>25kg/m^2 who were deemed insulin-resistant by the hyperinsulinemic -euglycemic clamp (with M/I value under median for men and women separately)

SUMMARY:
People who are overweight and/or obese are at risk of insulin resistance and type 2 diabetes. However, research has shown that some overweight and/or obese individuals remain insulin-sensitive and metabolically healthy despite their unhealthy body weight.

The investigators hypothesise that overweight and/or obese people who were deemed insulin-sensitive in previous studies will maintain their insulin sensitivity and metabolic health over time. The investigators also hypothesise that the preservation of insulin sensitivity will be accompanied by key metabolic health markers.

DETAILED DESCRIPTION:
While obesity is a risk factor for metabolic disease, sub cohorts with obesity not complicated by the metabolic syndrome have been described. These so called "metabolically healthy obese" may have reduced risk of type 2 diabetes, cardiovascular disease and all-cause mortality compared with individuals with obesity who present with components of the metabolic syndrome.

Longitudinal studies with diabetes and cardiovascular disease risk endpoints reported that individuals with obesity who are metabolically healthy (MHO) held an intermediate health status, such that they were still worse off than the healthy normal-weight individuals. While there have been studies evaluating the stability of the MHO phenotype over time, no study has reported the durability of insulin-sensitivity per se, as measured by the gold-standard hyperinsulinaemic-euglycaemic clamp. In the present study, we aimed to trace the change in insulin resistance/sensitivity, and to uncover predictors of insulin resistance in older age. The secondary aims were to trace the change in body composition, fat distribution and metabolic markers over time in a well-phenotyped cohort studied approximately 5-6 years apart.

ELIGIBILITY:
Inclusion Criteria:

* Participation in two previous studies conducted at the Garvan Institute of Medical Research Clinical Research Facility (described in the other publications 1-3).
* Willingness to give written informed consent and willingness to participate in the study.

Exclusion Criteria:

* Pregnant and/or lactating women.

Ages: 26 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants of two previous separate studies performed at the Garvan Institute of Medical Research (Sydney, Australia) were contacted by postal mail to gauge interest in participating in this follow-up study. In the original studies, exclusion criteria included weight change greater than 2 kg in the preceding 6 months, self-reported regular exercise for periods longer than 60 min/week, treatment with medications known to affect insulin sensitivity or carbohydrate metabolism, known renal, cardiac, or liver disease and current cancer, planning pregnancy, consumption of more than 20 and 40 g/day alcohol for women and men, respectively, and smoking >10 cigarettes/day
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Greenfield, MBBS, PhD, Principal Investigator — Garvan Institute of Medical Research; Dorit Samocha-Bonet, MSc, PhD, Principal Investigator — Garvan Institute of Medical Research
Locations (1):
- Dorit Samocha-Bonet, Darlinghurst, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonks KT, Ng Y, Miller S, Coster AC, Samocha-Bonet D, Iseli TJ, Xu A, Patrick E, Yang JY, Junutula JR, Modrusan Z, Kolumam G, Stockli J, Chisholm DJ, James DE, Greenfield JR. Impaired Akt phosphorylation in insulin-resistant human muscle is accompanied by selective and heterogeneous downstream defects. Diabetologia. 2013 Apr;56(4):875-85. doi: 10.1007/s00125-012-2811-y. Epub 2013 Jan 24. PMID 23344726
- [Background] Heilbronn LK, Campbell LV, Xu A, Samocha-Bonet D. Metabolically protective cytokines adiponectin and fibroblast growth factor-21 are increased by acute overfeeding in healthy humans. PLoS One. 2013 Oct 18;8(10):e78864. doi: 10.1371/journal.pone.0078864. eCollection 2013. PMID 24205333
- [Background] Samocha-Bonet D, Campbell LV, Viardot A, Freund J, Tam CS, Greenfield JR, Heilbronn LK. A family history of type 2 diabetes increases risk factors associated with overfeeding. Diabetologia. 2010 Aug;53(8):1700-8. doi: 10.1007/s00125-010-1768-y. Epub 2010 May 12. PMID 20461357
- [Result] Tang A, Coster ACF, Tonks KT, Heilbronn LK, Pocock N, Purtell L, Govendir M, Blythe J, Zhang J, Xu A, Chisholm DJ, Johnson NA, Greenfield JR, Samocha-Bonet D. Longitudinal Changes in Insulin Resistance in Normal Weight, Overweight and Obese Individuals. J Clin Med. 2019 May 8;8(5):623. doi: 10.3390/jcm8050623. PMID 31071971

RESULTS

PARTICIPANT FLOW:
Groups:
- Lean/Normal Weight: Individuals with BMI < 25 kg/m^2
- Overweight/Obese Insulin-Sensitive: Individuals with BMI > 25 kg/m^2 were categorised as Overweight/Obese Insulin-Sensitive if their M/I value was above the median M/I value for each gender
- Overweight/Obese Insulin-Resistant: Individuals with BMI > 25 kg/m^2 were categorised as Overweight/Obese Insulin-Resistant if their M/I were below the median M/I value for each gender
Period: Overall Study
Arm/Group | Lean/Normal Weight | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Started (Individuals who participated in 2 previous studies performed at the Garvan Institute) | 17 | 20 | 20
Completed | 17 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overweight/Obese Insulin-Sensitive: Individuals with BMI>25 kg/m^2 who were deemed insulin-sensitive at the baseline study
- Overweight/Obese Insulin-Resistant: Individuals with BMI>25 kg/m^2 who were deemed insulin-resistant at the baseline study
- Total: Total of all reporting groups
Arm/Group | Lean/Normal Weight | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant | Total
Number analyzed (Participants) | 17 | 20 | 20 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (11.1) | 54.2 (10.7) | 63.4 (10.7) | 57.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 12 | 27
  Male | 11 | 11 | 8 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 16 | 19 | 19 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Australia | 17 | 20 | 20 | 99

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: The change in insulin sensitivity (as measured by M-value normalised to insulin from hyperinsulinemic-euglycemic clamp) was determined "Follow-up Value - Baseline Value" /"Time between measurements". There were 2 time points 6 years apart
Time Frame: 6 years
Population: The hyperinsulinemic-euglycemic clamp was performed in a sub-cohort of n=9, 10 and 16 participants who were normal-weight, overweight/obese insulin-sensitive and overweight/obese insulin-resistant, respectively
Measure: Median (Inter-Quartile Range); unit: micro mol/min/Kg/mU/L/year
Groups:
- Lean/Normal Weight: Individuals with BMI<25 kg/m2 at the baseline study
- Overweight/Obese Insulin-Sensitive: Individuals with BMI>25 kg/m2 who were deemed insulin-sensitive at the baseline study
- Overweight/Obese Insulin-Resistant: Individuals with BMI>25 kg/m2 who were deemed insulin-resistant at the baseline study
Arm/Group | Lean/Normal Weight | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Number analyzed (Participants) | 9 | 10 | 16
micro mol/min/Kg/mU/L/year | 0.0105 [-0.0202 to 0.0163] | -0.0076 [-0.0380 to 0.0073] | 0.0041 [-0.0022 to 0.0109]

2. Secondary Outcome: Body Mass Index
Description: Change in body mass index (BMI) was determined as "Follow-up Value - Baseline Value" /"Time between measurements". There were 2 time points 6 years apart
Time Frame: 6 years
Population: All individuals who were followed up after 6 years were analyzed
Measure: Median (Inter-Quartile Range); unit: kg/m^2/year
Arm/Group | Lean/Normal Weight | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Number analyzed (Participants) | 17 | 20 | 20
kg/m^2/year | 0.0526 [-0.0179 to 0.2842] | 0.0941 [-0.0762 to 0.3689] | 0.0088 [-0.1867 to 0.2309]

3. Secondary Outcome: Waist Circumference
Description: Change in waist circumference was determined as "Follow-up Value - Baseline Value" /"Time between measurements". There were 2 time points 6 years apart
Time Frame: 6 years
Population: All individuals who were followed up after 6 years were analyzed
Measure: Median (Inter-Quartile Range); unit: cm/year
Arm/Group | Lean/Normal Weight | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Number analyzed (Participants) | 17 | 20 | 20
cm/year | 0.5263 [-0.1924 to 1.2060] | 0.4894 [-0.6522 to 1.1917] | 0.0000 [-1.0812 to 0.6588]

4. Secondary Outcome: Body Fat Mass
Description: Body fat mass from dual-energy X-ray absorptiometry (DXA) change was determined as "Follow-up Value - Baseline Value" /"Time between measurements". There were 2 time points 6 years apart
Time Frame: 6 years
Population: DXA was performed in a sub-cohort of n=11, 11 and 19 in normal weight, overweight/obese insulin-sensitive and overweight/obese insulin-resistant participants, respectively
Measure: Median (Inter-Quartile Range); unit: % of total body mass/year
Groups:
- Lean: The Lean group included all individuals with BMI < 25 kg/m2
- Overweight/Obese Insulin-Sensitive: Those with BMI > 25 kg/m2 were categorised as Overweight/Obese Insulin-Sensitive if their M/I value was above the median M/I value for each gender
- Overweight/Obese Insulin-Resistant: Those with BMI > 25 kg/m2 were categorised as Overweight/Obese Insulin-Resistant if their M/I were below the median M/I value for each gender
Arm/Group | Lean | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Number analyzed (Participants) | 11 | 11 | 19
% of total body mass/year | 0.2281 [-0.2256 to 0.8134] | 0.3696 [0.1465 to 0.5812] | 0.3478 [-0.0303 to 0.5745]

5. Secondary Outcome: Body FFM
Description: Body fat-free mass (FFM) from DXA change was determined as "Follow-up Value - Baseline Value" /"Time between measurements". There were 2 time points 6 years apart
Time Frame: 6 years
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: kg/year
Arm/Group | Lean | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Number analyzed (Participants) | 11 | 11 | 19
kg/year | -0.0382 [-0.2930 to 0.0771] | -0.1786 [-0.3613 to 0.0333] | -0.4017 [-0.7577 to 0.0277]

6. Secondary Outcome: Visceral Fat Volume
Description: Abdominal visceral fat volume from DXA change was determined as "Follow-up Value - Baseline Value" /"Time between measurements". There were 2 time points 6 years apart
Time Frame: 6 years
Population: Visceral fat volume was available in n=11, 10 and 18 normal weight, overweight/obese insulin-sensitive and overweight/obese insulin-resistant participants who undergone a DXA measure due to technical reasons
Measure: Median (Inter-Quartile Range); unit: cm^3/year
Arm/Group | Lean | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Number analyzed (Participants) | 11 | 10 | 18
cm^3/year | 13.3962 [-2.3225 to 75.3947] | 47.3351 [-12.6000 to 94.9231] | 46.2974 [27.1212 to 113.1915]

7. Secondary Outcome: Systolic Blood Pressure
Description: Change in Systolic Blood Pressure was determined as "Follow-up Value - Baseline Value" /"Time between measurements". There were 2 time points 6 years apart
Time Frame: 6 years
Population: All individuals who were followed up after 6 years were analyzed
Measure: Median (Inter-Quartile Range); unit: mmHg/year
Arm/Group | Lean | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Number analyzed (Participants) | 17 | 20 | 20
mmHg/year | 0.3704 [-0.3548 to 2.8373] | 0.9483 [-1.2137 to 2.5466] | 1.3593 [-0.1087 to 4.1122]

8. Secondary Outcome: Diastolic Blood Pressure
Description: Change in Diastolic Blood Pressure was determined as "Follow-up Value - Baseline Value" /"Time between measurements". There were 2 time points 6 years apart
Time Frame: 6 years
Population: All individuals who were followed up after 6 years were analyzed
Measure: Median (Inter-Quartile Range); unit: mmHg/year
Arm/Group | Lean | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Number analyzed (Participants) | 17 | 20 | 20
mmHg/year | 1.1290 [-0.3792 to 2.8535] | 0.4117 [-0.1567 to 1.3193] | 0.5662 [-0.3191 to 1.9224]

9. Secondary Outcome: Fasting Blood Glucose
Description: Change in fasting blood glucose was determined as "Follow-up Value - Baseline Value" /"Time between measurements". There were 2 time points 6 years apart
Time Frame: 6 years
Population: Fasting blood glucose concentration measure was available in a sub-cohort of n=16, 18 and 19 in normal weight, overweight/obese insulin-sensitive and overweight/obese insulin-resistant participants, respectively
Measure: Median (Inter-Quartile Range); unit: mmol/L/year
Arm/Group | Lean | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Number analyzed (Participants) | 16 | 18 | 19
mmol/L/year | -0.0151 [-0.0429 to 0.0500] | 0.0062 [-0.0333 to 0.0373] | -0.0254 [-0.0962 to 0.0512]

10. Secondary Outcome: Fasting Serum Insulin
Description: Change in fasting serum insulin was determined as "Follow-up Value - Baseline Value" /"Time between measurements". There were 2 time points 6 years apart
Time Frame: 6 years
Population: Fasting serum insulin measurement was available in a sub-cohort of n=16, 18 and 19 in normal weight, overweight/obese insulin-sensitive and overweight/obese insulin-resistant participants, respectively
Measure: Median (Inter-Quartile Range); unit: mU/L/year
Arm/Group | Lean | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
Number analyzed (Participants) | 16 | 18 | 19
mU/L/year | 0.2223 [-0.7104 to 1.2940] | 0.0855 [-0.6545 to 0.4863] | -0.2370 [-1.8802 to 0.5054]

ADVERSE EVENTS:
Time Frame: Serious and other [non-serious] adverse events were not collected or assessed as part of the study (observational study, no intervention administered)
Description: Not applicable (see above)
Groups:
- Lean/Normal Weight: Individuals with BMI < 25 kg/m2
Arm/Group | Lean/Normal Weight | Overweight/Obese Insulin-Sensitive | Overweight/Obese Insulin-Resistant
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study is limited by the small sample size, and the potential bias relating to populations likely to volunteer to studies which may have affected the findings. Furthermore, some data were missing for some individuals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes